CLINICAL TRIAL: NCT00869999
Title: Everolimus in Combination With Rituximab for Relapsed/Refractory Diffuse Large B Cell Lymphoma
Brief Title: Everolimus Plus Rituximab for Relapsed/Refractory Diffuse Large B Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Dana-Farber Cancer Institute (Other); Novartis (Industry)
Responsible Party: Principal Investigator, Jeremy Abramson, MD, Director, Lymphoma Program, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-002
Record Dates: First submitted 2009-03-25; First posted 2009-03-26 (Estimated); Results first posted 2014-10-27 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2013-10

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: rituximab; everolimus; DLBCL; mTOR
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Everolimus; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Everolimus — Taken orally once daily in the morning
Drug: rituximab — Given intravenously on Days 1, 8, 15, and 22 of Cycle 1 then on Day 1 of cycles 2-6

SUMMARY:
Everolimus is an oral mTOR inhibitor with demonstrated preliminary efficacy and safety in diffuse large B-cell lymphoma (DLBCL) in both preclinical and clinical studies. The purpose of this research study is to determine whether Everolimus plus rituximab is safe and effective in participants with relapsed or refractory DLBCL. Everolimus is an investigational drug that works by blocking a special protein that helps cancer cells grow. The safety and effectiveness of Everolimus in the treatment of DLBCL has not yet been fully determined and is still investigational. The other drug in this study, rituximab, is approved by the US Food and Drug Administration (FDA) for use in patients who have diffuse large B-cell lymphoma and certain other types of non-Hodgkin lymphoma. Rituximab is a drug that destroys both normal and cancerous B-cells.

DETAILED DESCRIPTION:
Participants will receive oral Everolimus and intravenous rituximab for DLBCL that has relapsed or been refractory to prior therapy.

* Each treatment cycle lasts 28 days (4 weeks). Everolimus will be taken orally, once daily in the morning.
* Rituximab will be administered by an intravenous (IV) infusion on Days 1, 8, 15 and 22 of Cycle 1. In Cycles 2-6, rituximab will be administered only on Day 1 of each cycle.
* Participants will come into the clinic weekly during the first cycle, then on Day 1 of all cycles thereafter. The following tests and procedures will be performed:
* Weekly During Cycle 1: blood tests
* Day 1 of all Subsequent Cycles: brief physical examination; review of current medications, treatments, symptoms and side effects; vital signs; performance status evaluation; blood tests.
* A full body CT and PET scan to assess the participants tumor will be done within 7 days of completing cycles 2, 4, 6, 9 and 12.

Responding subjects may receive up to 6 cycles of Everolimus plus rituximab, and an additional 6 months of oral Everolimus for participants continuing to respond.

ELIGIBILITY:
Inclusion Criteria:

* Histologically determined DLBCL that is relapsed or primary refractory after initial therapy
* Greater than 1 prior line of chemotherapy (including an anthracycline unless contraindicated) or immunotherapy. Patients must have relapsed after autologous stem cell transplantation, not be eligible for autologous stem call transplantation in the judgment of the investigator, or refuse autologous stem cell transplantation. Salvage chemotherapy and high dose conditioning for autologous stem cell transplantation count as two separate regimens.
* Measurable disease that has not been previously irradiated on PET-CT of at least 2cm, OR if the patient has had previous radiation to the marker lesion(s), there must be evidence of progression since the radiation. Imaging must be completed no greater than 3 weeks from study enrollment.
* ECOG performance status 0-2
* 18 years of age or older
* Life expectancy of greater than 3 months
* Adequate Organ and marrow function
* Fasting serum cholesterol of 300 mg/dl or less OR 7.75 mmol/L or less AND fasting triglycerides 2.5 x ULN or less

Exclusion Criteria:

* Currently receiving anticancer therapies or who have received anticancer therapies within 3 weeks of the start of the study drug
* Receiving any other investigational agents, or have received investigational agents within 4 weeks of beginning treatment
* Major surgery or significant traumatic injury within 4 weeks of start of study drug, patients who have not recovered from the side effects of any major surgery (defined as requiring general anesthesia) or patients that may require major surgery during the course of the study
* Known leptomeningeal or brain metastases. Imaging or spinal fluid analysis to exclude CNS involvement is not required, unless there is clinical suspicion by the treating investigator
* Known HIV infection
* Systemic fungal, bacterial, viral, or other infection not controlled
* Prior history of malignancy (except for non-melanoma skin cancer or in situ cervical or breast cancer) unless disease free for at least one year. Patients with prostate cancer are allowed if PSA is less than 1
* Patients should not receive immunization with attenuated live vaccines within one week of study entry or during study period
* Severely impaired lung function defined as DLCO of <60%
* Uncontrolled diabetes as defined by fasting serum glucose > 1.5 x ULN
* Liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of Everolimus
* Active bleeding diathesis
* Female patients who are pregnant or breastfeeding, or adults of reproductive potential who are not using effective birth control methods
* Prior treatment with an mTOR inhibitor
* Known hypersensitivity to murine antibodies,everolimus,other rapamycin
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study
* No chronic treatment with systemic corticosteroids or other immunosuppressive agents. Topical or inhaled corticosteroids are permitted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2009-05; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy S. Abramson, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconsess Medical Center, Boston, Massachusetts

REFERENCES:
- [Derived] Barnes JA, Jacobsen E, Feng Y, Freedman A, Hochberg EP, LaCasce AS, Armand P, Joyce R, Sohani AR, Rodig SJ, Neuberg D, Fisher DC, Abramson JS. Everolimus in combination with rituximab induces complete responses in heavily pretreated diffuse large B-cell lymphoma. Haematologica. 2013 Apr;98(4):615-9. doi: 10.3324/haematol.2012.075184. Epub 2012 Nov 9. PMID 23144193

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited in the lymphoma programs of the Massachusetts General Hospital Cancer Center, Dana-Farber Cancer Institute and Beth-Israel Deaconess Medical Center
Groups:
- Everolimus-Rituximab: All patients received treatment with everolimus-rituximab on this single am study. Everloimus was administered at a dose of 10mg by mouth once daily on days 1-28 of a 28-day cycle. Rituximab was administered at a dose of 375 mg/m3 intravenously weekly for four doses during cycle 1, and then on day 1 of cycles 2-6. After cycle 6, patients could receive an additional 6 months of everolimus monotherapy in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Everolimus-Rituximab
Started | 26
Completed | 24
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — removed prior to starting therapy | 1

BASELINE CHARACTERISTICS:
Population: 26 patients enrolled, 24 evaluable
Groups:
- Treatment Arm: All patients received treatment with everolimus-rituximab on this single am study
Arm/Group | Treatment Arm
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Secondary Outcome: Duration of Overall Response
Description: Duration of overall response is measured from the time measurement criteria are met for complete response or partial response until the first date that recurrent or progressive disease is objectively documented.
Time Frame: 2 years
Measure: Median (90% Confidence Interval); unit: months
Groups:
- Everolimus/Rituximab: All patients received treatment with everolimus-rituximab on this single am study. Everloimus was administered at a dose of 10mg by mouth once daily on days 1-28 of a 28-day cycle. Rituximab was administered at a dose of 375 mg/m3 intravenously weekly for four doses during cycle 1, and then on day 1 of cycles 2-6. After cycle 6, patients could receive an additional 6 months of everolimus monotherapy in the absence of disease progression or unacceptable toxicity.
Arm/Group | Everolimus/Rituximab
Number analyzed (Participants) | 24
months | 8.1 [4.9 to 16.3]

2. Secondary Outcome: Progression-free Survival
Description: Progression-free survival is defined as the duration of time from start of treatment to time of documentation of progression or death
Time Frame: 2 years
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Everolimus/Rituximab
Number analyzed (Participants) | 24
months | 2.9 [1.8 to 3.8]

3. Primary Outcome: Overall Response Rate
Description: Complete response plus partial response after 6 cycles. Response rate will be evaluated by using the modified Cheson criteria for lymphoma response. Complete response requires all of the following: 1) PET positive prior to therapy: mass of any size permitted if PET negative. Variable FDG-avid or PET negative prior to therapy: regression to normal size on CT (</= 1.5cm in their greatest transverse diameter for nodes >/= 1.5 cm before therapy) 2) Spleen (if enlarged before therapy) must have regressed in size and must not be palpable, 3) If bone marrow is known to be involved, repeat biopsy documents clearance. Partial response requires 1) >/= 50% decrease in SPD, 2) No new sites of disease or increase in the size of other nodes, liver or spleen, 3) Splenic and hepatic nodules must regress by at least 50% in SPD
Time Frame: Assessed at the conclusion of cycle 2, cycle 4 and cycle 6
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Everolimus/Rituximab
Number analyzed (Participants) | 24
percentage of participants | 38 [21 to 56]

ADVERSE EVENTS:
Arm/Group | Everolimus/Rituximab
Serious Adverse Events (participants affected / at risk) | 6/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Everolimus/Rituximab (N=24)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Viral hepatitis (Gastrointestinal disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus/Rituximab (N=24)
Fatigue (General disorders) | 8
Anorexia (General disorders) | 3
Rash (General disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 9
Anemia (Blood and lymphatic system disorders) | 10
Thrombocytopenia (Blood and lymphatic system disorders) | 11
Leukocytosis (Blood and lymphatic system disorders) | 8
Hyperglycemia (Metabolism and nutrition disorders) | 6
Hypertriglyceridemia (Metabolism and nutrition disorders) | 6
Infection with < grade 3 neutropenia (Infections and infestations) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No